CLINICAL TRIAL: NCT03555396
Title: A Couple-based Antiretroviral Therapy Adherence Intervention for People Who Inject Drugs in Kazakhstan
Brief Title: Couples ART Adherence Intervention for PWID in Kazakhstan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Alissa Davis, Professor of Social Work, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAR7144; 1K01DA044853-01A1 (NIH)
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-09

CONDITIONS: HIV Infections; Substance Use Disorders
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Subjects will receive an intervention is based off of current evidence-based practices and will consist of activities designed to strengthen support within the couple to improve adherence to antiretroviral therapy.
  Interventions: Behavioral: SMART Couples 2
- Standard of Care (Active Comparator): Standard of Care is the comparison arm that consists of care currently provided at the AIDS Center. Subjects will receive a consultation with a healthcare provider every three months, prescription refills, and blood draws for viral load and CD4 testing.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: SMART Couples 2 — The intervention will consist of 4 sessions with activities designed to strengthen communication and support within the couple to improve adherence to antiretroviral therapy and increase linkage to drug treatment services. The activities are based on cognitive-behavioral therapy. Participants' adherence will be monitored continuously through electronic monitoring devices and surveys completed at baseline and follow-up periods.
  Arms: Intervention
Behavioral: Standard of Care — Standard of Care consists of an appointment with an AIDS Center nurse at baseline and two months later. Under current Standard of Care in Almaty, no behavioral intervention is provided. Participants obtain prescription refills and give blood for viral load and CD4 tests once every 6 months.
  Arms: Standard of Care

SUMMARY:
The fastest growing HIV epidemics globally are driven by injection drug use, but only a small percentage of HIV-positive people who inject drugs (PWID) have achieved viral suppression. The proposed project will adapt a couple-based antiretroviral therapy (ART) adherence intervention for PWID and assess the feasibility and acceptability of conducting dried blood spot testing to objectively measure ART adherence as part of an intervention in a clinical setting. This project advances HIV intervention science by providing an intervention that leverages social support within the dyad to improve ART adherence among PWID, which could lead to increased viral suppression, thus decreasing HIV transmission and HIV-related morbidity and mortality.

DETAILED DESCRIPTION:
The purpose of this Mentored Research Scientist Development Award (K01) is to provide the candidate with the training and expertise needed to transition to research independence in the science of HIV prevention and intervention. The fastest growing HIV epidemics globally are driven by injection drug use. Central Asia has some of the highest rates of injection drug use and one of the fastest growing HIV epidemics in the world. HIV-positive people who inject drugs (PWID) face many barriers to antiretroviral therapy (ART) adherence, such as misperceptions about ART, stigma and substance use. Previous research among this population has shown that couple-based HIV interventions are highly efficacious at reducing risk behaviors, but there is currently no couple-based ART adherence intervention for PWID. The research aims of this proposal are to 1) identify core components of the SMART Couples intervention and other existing ART adherence intervention strategies and assess their appropriateness and feasibility as an integrated, couple-based ART adherence intervention for HIV+ PWID living in Kazakhstan (Phase 1); 2) adapt and refine SMART Couples and identify augmentative intervention strategies to create an integrated, couple-based ART adherence intervention for HIV+ PWID and their primary sex partners using results from Aim 1 (Phase 2); and 3a) pilot test the resulting couple-based intervention among 66 heterosexual PWID couples in Kazakhstan through a randomized control trial to assess the safety, feasibility, and acceptability of the intervention and obtain preliminary estimates of adherence outcomes in the intervention arm versus standard of care; and 3b) assess the feasibility and acceptability of conducting dried blood spot testing as part of an adherence intervention in a clinical setting (Phase 3). The proposed career development plan has been designed to augment the candidate's current training in epidemiology and enable her to 1) gain research skills in the design and adaptation of HIV interventions, with an emphasis on adherence among marginalized populations; 2) obtain methodological expertise in dyad and intensive longitudinal analysis and the triangulation of behavioral, biomedical, and technological data, particularly for the purposes of interpreting and analyzing these types of data to assess intervention efficacy and measure ART adherence; 3) acquire training in the conduct and analysis of qualitative in-depth interviews and focus groups, particularly for designing and adapting HIV interventions and assessing intervention feasibility and acceptability; and 4) increase professional skills for a successful independent research career. These training goals will be achieved through a combination of didactic courses, specialized workshops and seminars, hands-on research, and an interdisciplinary team of experts. The research findings and methodological skills to be gained from this K01 have wide applicability for disease research and high transferability across diverse research settings.

ELIGIBILITY:
Participant inclusion criteria for Phase 3: 66 couples (n=132) will participate in a randomized control trial of the adapted couple-based intervention.

Couples are eligible to participate if:

1. both partners are ≥18 years old,
2. both identify each other as their primary sexual partner (e.g. spouse, girlfriend/boyfriend, regular sexual partner),
3. the relationship has existed at least 3 months,
4. both report feeling safe participating with their partner in the study,
5. neither reports any severe physical or sexual violence perpetrated by the other partner in the past year,
6. both are able to provide informed consent and follow study procedures, and
7. both are fluent in Russian.

In addition, the "index case" (partner initially recruited from AIDS Center) must: (1) be confirmed HIV+ by the AIDS Center, (2) have been on ART at least 3 months, (3) not be virally suppressed according to the AIDS Center standard (<500 copies/ml), and (4) report injecting any drug in the past year.

Participant exclusion criteria for Phase 3:

Individuals who do not meet inclusion criteria or who meet any of the following criteria will be excluded from the study:

1. unable to provide informed consent,
2. unwilling or unable to participate in study procedures,
3. any condition that, in the opinion of the principal investigator and research staff, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alissa Davis, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Global Health Research Center of Central Asia, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
Unidentified data can be shared with other researchers in accordance with IRB regulations upon completion and analysis of the study.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available to other researchers starting 12 months after publication of the final results.
Access Criteria: Data can be accessed by emailing the PI of the study and obtaining appropriate Institutional Review Board (IRB) approvals.

REFERENCES:
- [Derived] Davis A, Rozental E, Bolger N, Gulyayev V, Gulyayev P, Denebayeva A, Wen H, Cui J, Terlikbayeva A, Primbetova S, Samandas J, Altice FL, Remien RH, Mergenova G. A Dyad-Based Intervention to Improve Adherence to Antiretroviral Therapy among People with HIV who Inject Drugs in Kazakhstan: Results of a Randomized Controlled Trial. AIDS Behav. 2026 Jan;30(1):1-13. doi: 10.1007/s10461-025-04841-5. Epub 2025 Aug 7. PMID 40773102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Almaty City AIDS Center from October 2020 to March 2023.
Pre-assignment Details: Participants were randomized as a dyad to the intervention or standard of care arm. Numbers reported represent individual participants (not dyads).
Groups:
- Intervention: Subjects will receive an intervention based off of current evidence-based practices that will consist of activities designed to strengthen support within the couple to improve adherence to antiretroviral therapy.
  SMART Couples 2: The intervention will consist of 3 sessions with activities designed to strengthen communication and support within the couple to improve adherence to antiretroviral therapy and increase linkage to drug treatment services. The activities are based on cognitive-behavioral therapy. Participants' adherence will be monitored continuously through electronic monitoring devices and surveys completed at baseline and follow-up periods.
Period: Overall Study
Arm/Group | Intervention | Standard of Care
Started | 64 | 68
Index Case | 32 | 34
Treatment Support Partner | 32 | 34
Completed | 61 | 65
Not Completed | 3 | 3
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Population: Each arm contained HIV-positive people who inject drugs and their treatment support partners. Treatment support partners may or may not be HIV-positive and may or may not inject drugs.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Standard of Care | Total
Number analyzed (Participants) | 64 | 68 | 132
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.11 (11.10) | 43.97 (9.59) | 45.01 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 31 | 59
  Male | 36 | 37 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 64 | 68 | 132
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 16 | 23 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 48 | 45 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Kazakhstan | 64 | 68 | 132
HIV status [Count of Participants; unit: Participants]
  HIV-positive | 45 | 50 | 95
  HIV-negative | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Adherence Rate to Antiretroviral Therapy
Description: Adherence rate is defined as the number of days the electronic pill bottle was opened to take medication (out of a total of 180 days).
Time Frame: Day 1 to Day 180 (daily)
Population: Participants analyzed included only those who were HIV-positive and who used the electronic monitoring device: 35 out of 64 in the intervention arm and 45 out of 68 in the standard of care arm. Not all participants were able to collect evaluable data using the device since there were no in-person study visits during the pandemic to help with troubleshooting.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 35 | 45
Days | 10.49 (11.21) | 14.02 (27.97)
Statistical Analysis 1: Comparison: Intervention vs Standard of Care; Test type: Superiority; p = 0.483, t-test, 2 sided; Mean Difference (Final Values) = -3.54, 95% CI 2-sided [-13.53 to 6.46]

2. Secondary Outcome: Number of Participants Stratified by Viral Load Suppression
Description: HIV viral load suppression was considered at ≤500 copies/ml in accordance with the Almaty AIDS Center testing standard. Participants were classified as virally suppressed or not based on their most recent viral load test result (at baseline and at the 6 month follow-up) obtained from electronic medical records at the AIDS Center.
Time Frame: 6 month follow-up
Population: Participants who had viral load testing data from the AIDS Center.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 40 | 40
Participants
  Detectable viral load (>500 copies/ml) at baseline decreased to virally suppressed at 6 months | 14 | 11
  Viral load remained detectable (>500 copies/ml) at baseline and 6 months | 12 | 11
  Viral load remained suppressed (≤500 copies/ml) at baseline and 6 months | 14 | 18
Statistical Analysis 1: Comparison: Intervention vs Standard of Care; Test type: Superiority; p = 0.637, Chi-squared

3. Secondary Outcome: Medication Adherence Rate (Self-Report Score)
Description: Self-reported; 3 item scale (Self-Report Measure for Medication Adherence by Wilson et al., AIDS & Behavior, 2016) asking participants how well they took their medication in the past 30 days (average score on a 0-100 scale). 0 = low adherence and 100 = high adherence.
Time Frame: 6 month follow-up
Population: Only HIV-positive participants had outcome data in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 45 | 50
units on a scale
  Baseline | 69.29 (2.52) | 68.33 (2.20)
  6-month follow-up | 86.73 (2.56) | 76.23 (2.37)
Statistical Analysis 1: Comparison: Intervention vs Standard of Care; Test type: Superiority; p = 0.037, Mixed Models Analysis — Difference in mean change in adherence from baseline to 6 month follow-up between individuals in the intervention and control arms; Multilevel linear mixed model with random effects (dyad & intercept); adjusting for participant age, sex, baseline adherence, and partner HIV status; Mean Difference (Net) = 9.54, 95% CI 2-sided [0.59 to 18.49]

4. Secondary Outcome: Number of Subjects That Had Access to Substance Use Treatment
Description: Self-reported; participants reported if they were currently receiving methadone or opioid substitution therapy
Time Frame: 6 month follow-up
Population: Only participants who reported ever injecting drugs who completed the 6-month follow-up survey: 42 out of 64 in the intervention arm and 49 out of 68 in the standard of care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Standard of Care
Number analyzed (Participants) | 42 | 49
Participants | 1 | 3
Statistical Analysis 1: Comparison: Intervention vs Standard of Care; Test type: Superiority; p = 0.621, Chi-squared; Fisher's Exact Test used for small sample sizes

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Intervention | Standard of Care
All-Cause Mortality (participants affected / at risk) | 3/64 | 1/68
Serious Adverse Events (participants affected / at risk) | 4/64 | 3/68
Other Adverse Events (participants affected / at risk) | 3/64 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=64) | Standard of Care (N=68)
Hospitalization (Infections and infestations) | 4 (4) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=64) | Standard of Care (N=68)
Jailed (Social circumstances) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Data were collected during the Coronavirus-19 (COVID-19) pandemic. Many participants experienced problems using electronic monitoring devices, and research staff were not allowed to make home visits to trouble-shoot. During COVID-19, many opioid substitution therapy (OST) clinics in Kazakhstan also closed, making it difficult for participants to access (OST).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/96/NCT03555396/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT03555396/SAP_001.pdf